CLINICAL TRIAL: NCT04151303
Title: The Optimal Timing for Cerclage Removal
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yaniv Zipori MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0410-19-RMB
Record Dates: First submitted 2019-07-02; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Disease of A Newborn
Keywords: RDS; CERCLAGE; CERVIX INSUFFICIENCY
MeSH Terms: interventions — Cerclage, Cervical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cerclage 1: Time to delivery after cerclage removal Between 36-36.6 weeks' gestation - group 1
  Interventions: Procedure: Cervical cerclage
- Cerclage 2: Time to delivery after cerclage removal Between 37-37.6 weeks' gestation - group 2
  Interventions: Procedure: Cervical cerclage
- Cerclage 3: Between 38-38.6 weeks' gestation - group 3
  Interventions: Procedure: Cervical cerclage
- Cerclage 4: Time to delivery after cerclage removal Beyond 39 weeks' gestation - group 4
  Interventions: Procedure: Cervical cerclage

INTERVENTIONS:
Procedure: Cervical cerclage — Cervical cerclage and cervical cerclage removal

SUMMARY:
Women with a history of cervical insufficiency can be managed with elective cervical cerclage placed at the beginning of the second trimester. The McDonald technique is the most commonly used. Though lack a robust scientific evidence, the cerclage is removed electively at 36-37 weeks of gestation in order to avoid maternal cervical laceration. In addition, the incidence of spontaneous delivery is nearly 20% within 72 hours after ceclage removal, thus elective cerclage removal at 36-37 weeks may also put the newborns at complications associated with iatrogenic late preterm/early term delivery

DETAILED DESCRIPTION:
The optimal timing of cervical cerclage removal is yet unclear.

In the present study we will evaluate maternal and neonatal outcome variables after elective removal of the cerclage, and may suggest a gestational week cut-off for optimal cerclage removal/

Primary outcome:

Neonatal respiratory morbidity after cerclage removal. The respiratory outcome will be compared across each gestational week of delivery after cerclage removal, that is; group 1 (36-36.6 weeks), group 2 (37-37.6 weeks), group 3 (38-38.6 weeks), group 4 (beyond 39 weeks).

Secondary outcomes:

Time interval between cerclage removal and gestational age of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Elective or emergent cerclage in the current pregnancy
* Cerclage that was removed after 36 weeks of pregnancy

Exclusion Criteria:

* Multiple pregnancies
* Major congenital anomalies
* Cerclage removal before 36weeks of pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: - Women with singleton pregnancies with elective or emergent cerclage that was electively removed after 36 weeks of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Cercalge removal and neonatal morbidity | 1 year
  Neonatal respiratory morbidity after cerclage removal

SECONDARY OUTCOMES:
The optimal timing for cerclage removal | 1 year
  Time interval between cerclage removal and gestational age of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Zipori, M.D, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Yet undecided